CLINICAL TRIAL: NCT06653816
Title: Comparing the New Exponential Injury Severity Score (EISS) with the Injury Severity Score (ISS) and the New Injury Severity Score (NISS) in Polytrauma Patients for Survival Prediction and ICU Admission in Assiut University Hospitals
Brief Title: Comparing Exponential Injury Severity Score (EISS) with Injury Severity Score (ISS) and New Injury Severity Score (NISS)
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Mohamed Moussa, Principal Investigator, Assiut University
Other Study IDs: EISS-NISS-ISS
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Polytrauma
Keywords: EISS; NISS; ISS
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Trauma is defined as a physical injury from an external source of sudden onset and severity, which require immediate medical attention. Polytrauma is a short verbal equivalent commonly used for severely injured patients usually with associated injury (i.e., two or more severe injuries in at least two different areas of the body), less often with a multiple injury (i.e., two or more severe injuries in one body area). Polytrauma patients usually have a much higher risk of mortalities and disabilities than the risk of expected mortalities in individual injuries patients.

Despite improvements in trauma systems worldwide, trauma continues to be one of the leading causes of death and disability in all age groups, especially the young and middle age group. Approximately 5.8 million people die each year due to trauma related injuries, representing 8% of the worldwide mortality.

For studying the outcomes of trauma, accurate and reliable methodological tools are required for appropriate scoring of severity and outcome prediction.

Trauma scores were designed to facilitate the triage of patients in the Emergency Room (ER) and identify patients with Polytrauma with low chances of survival. Those scores were meant to organize and improve the quality of trauma care systems, and to assess resources allocation.

Trauma patients present to the emergency department (ED) with a great variety of injuries and diseases. To address these, the Abbreviated Injury Scale (AIS) system defines the severity of injury throughout the different regions of the body. It is an anatomically based, consensus derived, global severity scoring system that classifies an individual injury by body region according to its relative severity on a 6-point scale (1 = minor and 6 = maximal). The system is constantly revised, expanded, and improved, and the Association for the Advancement of Automotive Medicine recently announced its latest revision, the AIS 2005-Update 2008 and AIS 2015. To summarize a single patient's multiple injures into a single score, the Injury Severity Score (ISS) was created by Baker et al. in 1974, which has been considered the "gold standard" among anatomic injury severity indicators. It is based on the AIS severity values, that is, the summation of the squares of the severity digit in the AIS of the most severe injuries, in three of six predefined body regions.

However, the ISS only includes one injury in each body region, which leads to possible inclusion of a less severe injury in other body regions rather than another serious injury in the same body region. To overcome this limitation, a modified ISS, the New Injury Severity Score (NISS) was introduced by Osler et al. in 1997. NISS is simply the sum of squares of the three most severe injuries, regardless of the body regions injured.

Further, Wang et al. have created the Exponential Injury Severity Score (EISS) in 2014 by modifying the AIS system. The EISS was computed as the simple change in AIS values by raising each AIS severity score (1-6) by 3 taking a power of AIS minus 2, and then summing the three most severe scores (i.e., highest AIS values), regardless of body regions. With this exponential transformation of the AIS values, the EISS is expected to be more reflective of the true severity of injuries in a patient with polytrauma. In Wang's study, the EISS is reported to be more predictive of survival; therefore, it might be used as the standard summary measure of human trauma.

DETAILED DESCRIPTION:
Trauma is defined as a physical injury from an external source of sudden onset and severity, which require immediate medical attention. Polytrauma is a short verbal equivalent commonly used for severely injured patients usually with associated injury (i.e., two or more severe injuries in at least two different areas of the body), less often with a multiple injury (i.e., two or more severe injuries in one body area). Polytrauma patients usually have a much higher risk of mortalities and disabilities than the risk of expected mortalities in individual injuries patients.

Despite improvements in trauma systems worldwide, trauma continues to be one of the leading causes of death and disability in all age groups, especially the young and middle age group. Approximately 5.8 million people die each year due to trauma related injuries, representing 8% of the worldwide mortality.

Even though polytrauma can occur due to different causes such as road traffic accidents, fall from heights, bullet injuries, suicide, and homicide. Yet the leading cause of traumatic related causes of death worldwide is road traffic accidents. Egypt has experienced an alarming increase in the burden of traumatic injuries. In 2015, according to the World Health Organization, Egypt had one of the highest rates of road accidents worldwide, with more than 12,000 fatalities each year, one of the highest among Eastern Mediterranean Region (EMR) countries.

Although 90% of world's road trauma related fatalities occur in low- and middle-income countries, Injury prevention and trauma care programs in these countries have remained deficient.

For studying the outcomes of trauma, accurate and reliable methodological tools are required for appropriate scoring of severity and outcome prediction. Trauma scores were designed to facilitate the triage of patients in the Emergency Room (ER) and identify patients with Polytrauma with low chances of survival. Those scores were meant to organize and improve the quality of trauma care systems, and to assess resources allocation.

More than 50 scoring systems have been published for the classification of trauma patients in the field, emergency room, and intensive care settings. There are three main groups of trauma scores: Anatomical, Physiological, and Combined scores. Anatomical scores describe all the injuries recorded by clinical examination, imaging, surgery or autopsy and measure lesion severity {ex. Abbreviated Injury Scale (AIS) - Injury Severity Score (ISS) - New Injury Severity Score (NISS) -Organ Injury Scale (OIS) - Anatomic Profile -International Classification of Diseases (ICD-9) Injury Severity Score (ICISS)}. Physiological scores describe changes happened due to the trauma and translated by changes in vital signs and consciousness {ex. Revised Trauma Score - Glasgow Coma Score - APACHE scoring (Acute Physiology and Chronic Health Evaluation - (APACHE I, II, III) -Rapid Emergency Medicine Score (REMS)}. Combined scores include both anatomical and physiological criteria {ex. Trauma and Injury Severity Scores (TRISS) - A Severity Characterization of Trauma (ASCOT)-Kampala Trauma Score (KTS)}.

Trauma patients present to the emergency department (ED) with a great variety of injuries and diseases. To address these, the Abbreviated Injury Scale (AIS) system defines the severity of injury throughout the different regions of the body. It is an anatomically based, consensus derived, global severity scoring system that classifies an individual injury by body region according to its relative severity on a 6-point scale (1 = minor and 6 = maximal). The system is constantly revised, expanded, and improved, and the Association for the Advancement of Automotive Medicine recently announced its latest revision, the AIS 2005-Update 2008 and AIS 2015. To summarize a single patient's multiple injures into a single score, the Injury Severity Score (ISS) was created by Baker et al. in 1974, which has been considered the "gold standard" among anatomic injury severity indicators. It is based on the AIS severity values, that is, the summation of the squares of the severity digit in the AIS of the most severe injuries, in three of six predefined body regions.

However, the ISS only includes one injury in each body region, which leads to possible inclusion of a less severe injury in other body regions rather than another serious injury in the same body region. To overcome this limitation, a modified ISS, the New Injury Severity Score (NISS) was introduced by Osler et al. in 1997. NISS is simply the sum of squares of the three most severe injuries, regardless of the body regions injured.

Further, Wang et al. have created the Exponential Injury Severity Score (EISS) in 2014 by modifying the AIS system. The EISS was computed as the simple change in AIS values by raising each AIS severity score (1-6) by 3 taking a power of AIS minus 2, and then summing the three most severe scores (i.e., highest AIS values), regardless of body regions. With this exponential transformation of the AIS values, the EISS is expected to be more reflective of the true severity of injuries in a patient with polytrauma. In Wang's study, the EISS is reported to be more predictive of survival; therefore, it might be used as the standard summary measure of human trauma.

The aim of this study is to compare the ability of the new Exponential Injury Severity Score (EISS) with that of the Injury Severity Score (ISS) and the New Injury Severity Score (NISS) to identify patients at risk of in-hospital mortality or ICU admission and predict survival in Assiut University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

- traumatic patients with multiple trauma, both genders "without intently selected certain gender" and had 18 years old or more.

Exclusion Criteria:

* Patients who are less than 18 years old.
* Patients with end stage chronic disease .
* Patients with localized individual trauma will be excluded from this study.
* Patients refusing study .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: traumatic patients with multiple trauma of both genders "without intently selected certain gender" and had 18 years old or more.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 30 days
  Mortality "death" during the 30 day follow-up

SECONDARY OUTCOMES:
Rate of Intensive Care Unit admission | Day 0
  Admission to the Intensive Care Unit or High Dependency Unit from the Emergency Department
Rate of hospital admission | Day 0
  Admission to hospital from the Emergency Department
Rate of readmission in the Emergency Department | Hour 72, Day 30
  Re-visits to the Emergency Department after the index-visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuo SCH, Kuo PJ, Chen YC, Chien PC, Hsieh HY, Hsieh CH. Comparison of the new Exponential Injury Severity Score with the Injury Severity Score and the New Injury Severity Score in trauma patients: A cross-sectional study. PLoS One. 2017 Nov 9;12(11):e0187871. doi: 10.1371/journal.pone.0187871. eCollection 2017. PMID 29121653
- [Background] Wang MD, Fan WH, Qiu WS, Zhang ZL, Mo YN, Qiu F. The exponential function transforms the Abbreviated Injury Scale, which both improves accuracy and simplifies scoring. Eur J Trauma Emerg Surg. 2014 Jun;40(3):287-94. doi: 10.1007/s00068-013-0331-1. Epub 2013 Oct 5. PMID 26816062
- [Background] Osler T, Baker SP, Long W. A modification of the injury severity score that both improves accuracy and simplifies scoring. J Trauma. 1997 Dec;43(6):922-5; discussion 925-6. doi: 10.1097/00005373-199712000-00009. PMID 9420106
- [Background] Baker SP, O'Neill B, Haddon W Jr, Long WB. The injury severity score: a method for describing patients with multiple injuries and evaluating emergency care. J Trauma. 1974 Mar;14(3):187-96. No abstract available. PMID 4814394
- [Background] Beuran M, Negoi I, Paun S, Runcanu A, Gaspar B, Vartic M. [Trauma scores: a review of the literature]. Chirurgia (Bucur). 2012 May-Jun;107(3):291-7. Romanian. PMID 22844826
- [Background] Guzzo JL, Bochicchio GV, Napolitano LM, Malone DL, Meyer W, Scalea TM. Prediction of outcomes in trauma: anatomic or physiologic parameters? J Am Coll Surg. 2005 Dec;201(6):891-7. doi: 10.1016/j.jamcollsurg.2005.07.013. Epub 2005 Oct 13. PMID 16310692
- [Background] Elachi IC, Yongu WT, Odoyoh OO, Mue DD, Ogwuche EI, Ahachi CN. An epidemiological study of the burden of trauma in Makurdi, Nigeria. Int J Crit Illn Inj Sci. 2015 Apr-Jun;5(2):99-102. doi: 10.4103/2229-5151.158404. PMID 26157653
- [Background] Bikbov B, Perico N, Remuzzi G. Mortality landscape in the global burden of diseases, injuries and risk factors study. Eur J Intern Med. 2014 Jan;25(1):1-5. doi: 10.1016/j.ejim.2013.09.002. Epub 2013 Sep 29. PMID 24084027
- [Background] Marsden NJ, Tuma F. Polytraumatized Patient. 2023 Jul 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554426/ PMID 32119313
- [Background] Rau CS, Wu SC, Kuo PJ, Chen YC, Chien PC, Hsieh HY, Hsieh CH. Polytrauma Defined by the New Berlin Definition: A Validation Test Based on Propensity-Score Matching Approach. Int J Environ Res Public Health. 2017 Sep 11;14(9):1045. doi: 10.3390/ijerph14091045. PMID 28891977
- [Background] Cernea D, Novac M, Dragoescu PO, Stanculescu A, Duca L, Al-Enezy AA, Dragoescu NA. Polytrauma and Multiple Severity Scores. Curr Health Sci J. 2014 Oct-Dec;40(4):244-8. doi: 10.12865/CHSJ.40.04.02. Epub 2014 Dec 14. PMID 26793320
- [Background] Lendrum RA, Lockey DJ. Trauma system development. Anaesthesia. 2013 Jan;68 Suppl 1:30-9. doi: 10.1111/anae.12049. PMID 23210554
- See also: World Health Organization. Injuries and violence. Published March 19, 2021. — https://www.who.int/news-room/fact-sheets/detail/injuries-and-violence
- See also: The Global Road Safety Facility (GRSF), World Health Organization. Egypt's Road Safety Country Profile. Published 2016. — https://www.roadsafetyfacility.org/country/egypt